CLINICAL TRIAL: NCT00003946
Title: Phase II Study of Danazol in Advanced or Recurrent Endometrial Cancer
Brief Title: Danazol in Treating Patients With Advanced or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067139; GOG-0180
Record Dates: First submitted 1999-11-01; First posted 2004-06-25 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2004-07

CONDITIONS: Endometrial Cancer
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Danazol

INTERVENTIONS:
Drug: danazol

SUMMARY:
RATIONALE: Hormone therapy may be an effective treatment for endometrial cancer.

PURPOSE: Phase II trial to study the effectiveness of danazol in treating patients with advanced or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of danazol in patients with advanced or recurrent endometrial cancer. II. Determine the nature and toxicity of danazol in these patients.

OUTLINE: Patients receive oral danazol 4 times per day for at least 4 weeks. Patients with partial response, complete response, or stable disease continue treatment in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 23-56 patients will be accrued for this study within 26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced or recurrent endometrial cancer that is not amenable to curative surgery or radiotherapy Measurable disease Tumor at least 1.0 cm by 1.0 cm per x-ray or physical exam OR Tumor at least 2.0 cm by 2.0 cm per CT scan, MRI, or ultrasound

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3000/mm3 Platelet count at least 100,000/mm3 No history of porphyria Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 2 mg/dL Other: No concurrent or prior malignancy within past 5 years (except nonmelanoma skin cancer) or for which patient received chemotherapy Not pregnant or nursing Fertile patients must use effective contraception Must have tissue available for estrogen receptor/ progesterone receptor analysis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: At least 3 weeks since prior surgery and recovered

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Covens, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (73):
- United States (71):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Canada (2):
  - NCIC-Clinical Trials Group, Kingston, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario

REFERENCES:
- [Result] Covens A, Brunetto VL, Markman M, Orr JW, Lentz SS, Benda J; Gynecologic Oncology Group. Phase II trial of danazol in advanced, recurrent, or persistent endometrial cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2003 Jun;89(3):470-4. doi: 10.1016/s0090-8258(03)00149-5. PMID 12798713